CLINICAL TRIAL: NCT04643314
Title: Effect of Video-based Guided Self-reflection on Intraoperative Skills: a Pilot Randomized Controlled Trial
Brief Title: Effect of Video-based Guided Self-reflection on Intraoperative Skills
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Dr. Liane S. Feldman, Professor of Surgery and Chief of the Division of General Surgery at McGill University, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2020-6348
Record Dates: First submitted 2020-06-24; First posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Laparoscopy
Keywords: laparoscopic surgical skills; self-reflection; operative recording; laparoscopic cholecystectomy; surgical education

STUDY DESIGN:
Intervention Model Description: The study will be a parallel, two-groups, assessor-blind, single-center, pilot randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, the participants (resident trainees) cannot be blinded, however the assessors (attending surgeons) who will rate performance will be unaware of group allocation. Any inadvertent unblinding will be reported.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided video-based self-evaluation (Experimental): In addition to their usual residency training, participants randomized to this group will undergo the following interventions:
  The participants will be asked to review their own operating room recordings (of each of the 5 consecutive submitted laparoscopic cholecystectomy cases that the participant acted as the primary operator) and to assess themselves (within 72 hours (3 days) of the procedure) using validated intra-operative assessment tools. The completion of the self-evaluations is to guide and document video-based self-reflection. The duration of self-assessment/reflection session will be up do the participant. Residents in this group will have unlimited access to their recordings through the web-based platform. On the other hand, they will not be able to access the battery of assessment forms after the third day following the procedure.
  Interventions: Other: Guided video-based self-evaluation
- Traditional intraoperative teaching (No Intervention): Subjects randomized to this group will undergo their usual residency training.
  The recordings of the 5 submitted consecutive laparoscopic cholecystectomy procedures performed by the participant as the primary operator will be stored. However participants in this arm of the study will not have access to the uploaded videos until the end of the study.

INTERVENTIONS:
Other: Guided video-based self-evaluation — In addition to their usual residency training, participants randomized to this group will undergo the following interventions:
  The participants will be asked to review their own operating room recordings (of each of the 5 consecutive submitted laparoscopic cholecystectomy cases that the participant acted as the primary operator) and to assess themselves (within 72 hours (3 days) of the procedure) using validated intra-operative assessment tools. The completion of the self-evaluations is to guide and document video-based self-reflection. The duration of self-assessment/reflection session will be up do the participant. Residents in this group will have unlimited access to their recordings through the web-based platform. On the other hand, they will not be able to access the battery of assessment forms after the third day following the procedure.
  Arms: Guided video-based self-evaluation

SUMMARY:
While video-assisted structured feedback by expert surgeons significantly improves laparoscopic skill acquisition in surgical trainees, this method is resource intensive and may have limited feasibility outside of research settings. Self-assessment and reflection are integral parts of medical experiential learning; however the value of video-based self-reflection in enhancing surgical skill acquisition remains to be determined.

The objective of the proposed pilot study is to investigate the feasibility of conducting a full-scale randomized controlled trial (RCT) aimed to evaluate the effectiveness of coached video-based self-reflection approach on surgical trainee performance of laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
The study will be a parallel, two-groups, assessor-blind, single-center, pilot randomized controlled trial with participants (surgical trainees) individually allocated on a 1:1 ratio to intervention group (guided video-based self-evaluation in addition to traditional intraoperative teaching by faculty surgeons) and a control group (traditional intraoperative teaching alone).

All the trainees participating in this trial will be asked to submit intra-operative video-recordings of 5 consecutive laparoscopic cholecystectomies performed by them as the primary operator.

In this trial the intervention group participants will be asked to perform a guided self-assessment of their intra-operative skills by watching their operative video-recording. The trainee's self-assessment will be guided by validated intra-operative performance assessment tools. The control group will not have access to their recorded video submissions during the duration of this study.

Outcomes assessed will include trainee's intra-operative performance and time to completion of surgical procedure, Information generated from the pilot study will help inform a full-scale RCT by testing the study procedures. Feasibility outcomes will include number of trainees and surgeons approached, consented and randomized and adherence with intervention(surgeons: intra-operative assessments; trainees: video-based assessments). Data from this pilot study will inform the calculation of sample size requirements for the full-scale RCT.

ELIGIBILITY:
Inclusion Criteria:

* All residents involved at the McGill General Surgery Program (total of 35 residents on clinical rotations)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Rate of recruitment (acceptability of the trial by trainees) | 1 year
  % of eligible residents who agree to participate in the study
Feasibility: Rate of recruitment (acceptability of the trial by attending surgeons) | 1 year
  % of eligible attending surgeons who agree to participate in the study
Feasibility: Adherence to intervention | 1 year
  % of adherence with intervention (surgeons: intra-operative assessments; trainees: video-based assessments)
Feasibility: Rate of missing assessment data | 1 year
  % of missing responses

SECONDARY OUTCOMES:
Intraoperative performance- In-person: attending surgeon | 1 year
  Intra-operative performance will be assessed by the attending surgeon (present at time of the operation) after each operation (within 72 hours) using the following four tools:
  The Global Operative Assessment of Laparoscopic Skills (GOALS) Score 5-25 with higher score signifying better skills Operative Performance Rating System (OPRS) Score 10-50 with higher score signifying better skills Eubanks checklist 0-100% with higher score signifying better skills The O-SCORE Entrustability Scale 1-5 with higher score signifying better skills
Procedural times | 1 year
  Time to the following events:
  1. time to critical view of safety after completion of adhesiolysis,
  2. time to detachment of the gallbladder from the liver bed after division of the cystic artery and duct
  3. total procedure time (from insertion of first trocar to extraction of the gallbladder).
Perceived usefulness | through study completion, an average of 1 year
  all participants will be asked to evaluate the perceived utility of video-based self-reflection at baseline. This will be repeated at the end of the trial for the intervention group. In addition, they will be queried about the ease of executing the intervention (recording, storage and retrieval of their procedures) at the end of trial.
Mindset | through study completion, an average of 1 year
  Dweck Mindset instrument, DMI
Intraoperative performance-Video-based: blinded expert assessor | 1 year
  Intra-operative performance will be assessed by two expert assessors (MIS attending surgeons blinded to the case number or group allocation of the participants) using the following three tools:
  The Global Operative Assessment of Laparoscopic Skills (GOALS) Score 5-25 with higher score signifying better skills Operative Performance Rating System (OPRS) Score 10-50 with higher score signifying better skills Eubanks checklist 0-100% with higher score signifying better skills

CONTACTS AND LOCATIONS:
Overall Officials: Liane S Feldman, MD, Principal Investigator — McGill University
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be available to other researchers